CLINICAL TRIAL: NCT05109650
Title: A Phase 1, Multi-Center, Open-Label Study to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BAT6026 as Monotherapy and in Combination With BAT1308 in Patients With Advanced Solid Tumours
Brief Title: Assessment of Safety and Preliminary Efficacy With BAT6026 in Solid Tumour Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Considering that the high budget will affect the subsequent development, it is decided to terminate the test voluntarily
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-6026-002-CR
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumour
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 0.1mg/kg of BAT6026 + 300mg of BAT1308 (Experimental): 0.1mg/kg of BAT6026 Ⅳ infusions at cycle 1(monotherapy), and 0.1mg/kg of BAT6026 IV infusions + 300mg of BAT1308 IV infusions(combination therapy) from cycle 2 until end of treatment
  Interventions: Drug: BAT6026; Drug: BAT1308
- 0.3mg/kg of BAT6026 + 300mg of BAT1308 (Experimental): 0.3mg/kg of BAT6026 Ⅳ infusions at cycle 1(monotherapy), and 0.3mg/kg of BAT6026 IV infusions + 300mg of BAT1308 IV infusions(combination therapy) from cycle 2 until end of treatment
  Interventions: Drug: BAT6026; Drug: BAT1308
- 1mg/kg of BAT6026 + 300mg of BAT1308 (Experimental): 1mg/kg of BAT6026 Ⅳ infusions at cycle 1(monotherapy), and 1mg/kg of BAT6026 IV infusions + 300mg of BAT1308 IV infusions(combination therapy) from cycle 2 until end of treatment
  Interventions: Drug: BAT6026; Drug: BAT1308
- 3mg/kg of BAT6026 + 300mg of BAT1308 (Experimental): 3mg/kg of BAT6026 Ⅳ infusions at cycle 1(monotherapy), and 3mg/kg of BAT6026 IV infusions + 300mg of BAT1308 IV infusions(combination therapy) from cycle 2 until end of treatment
  Interventions: Drug: BAT6026; Drug: BAT1308
- 6mg/kg of BAT6026 + 300mg of BAT1308 (Experimental): 6mg/kg of BAT6026 Ⅳ infusions at cycle 1(monotherapy), and 6mg/kg of BAT6026 IV infusions + 300mg of BAT1308 IV infusions(combination therapy) from cycle 2 until end of treatment
  Interventions: Drug: BAT6026; Drug: BAT1308
- 10mg/kg of BAT6026 + 300mg of BAT1308 (Experimental): 10mg/kg of BAT6026 Ⅳ infusions at cycle 1(monotherapy), and 10mg/kg of BAT6026 IV infusions + 300mg of BAT1308 IV infusions(combination therapy) from cycle 2 until end of treatment
  Interventions: Drug: BAT6026; Drug: BAT1308

INTERVENTIONS:
Drug: BAT6026 — IV infusions
  Other Names: Recombinant Anti-OX40 Antibody Solution for Injection
Drug: BAT1308 — Ⅳ infusions
  Other Names: Recombinant Anti-PD-1 Antibody Solution for Injection

SUMMARY:
This is a multicenter, open-label, Phase 1 dose-escalation study of BAT6026, an OX40 monoclonal antibody, combined with the anti-PD-1 IgG4 monoclonal antibody BAT1308 in subjects with advanced solid tumours. After a screening period of up to 28 days, qualified subjects will be enrolled to receive their assigned dose regimen until disease progression or intolerable toxicity, withdrawal of consent, per Investigator decision, or end of study, whichever occurs first. The maximum treatment duration is 1 year. Subjects who remain on treatment in the absence of disease progression for more than 1 year may continue to receive study drug for the next cycle at the maximum of 2 years.

DETAILED DESCRIPTION:
Although the success of immune checkpoints like PD-1/PD-L1 and CTLA-4 has provided more alternatives and benefit to cancer patients, there are still much unmet need in tumour patients. That is why novel immunomodulatory drugs with other mechanisms of action still needed to be developed and tested clinically. OX40 is a co-stimulatory immune checkpoint which is contrary to PD-1 or CTLA4. Similar to other TNFSF members, three OX40 molecules were clustered when binding to one OX40L ligand on activated APCs. The clustered OX40s then directly activate NF-kB, PI3K/PKB and NFAT signal pathways to activate CD4+ and CD8+T cells 9. Thus, antibody targeting OX40 should be an agonist antibody which can be crosslinked by FcyR of effector cells. As the mechanism and signal pathways mediated by OX40 to activate T cells are different from those mediated by PD-1 and CTLA-4, targeting on OX40 may provide different clinical benefit for patients than treating with PD-1 and CTLA-4 therapies.

To enhance activation on T cells, combination treatment with PD-1, PD-L1, or CTLA-4 antibodies is a feasible approach for anti-OX40 immunotherapy. The effect of combination treatment of BAT6026 with an anti-PD1 antibody, BAT1308, in mouse tumour model was examined in the in vivo pharmacology study. MC38 murine colon carcinoma cells were inoculated in PD-1/OX40-dual-humanized mice.

Therefore, besides exploration as a monotherapy, finding a combination agent(s) and a suitable indication(s) would also be an encouraging direction for clinical development of BAT6026.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects able to give voluntary informed consent and understand the study and are willing to follow and complete all the test procedures.
* 2. Male or female, age ≥ 18 years.
* 3. Life expectancy ≥3 months.
* 4. ECOG performance status ≤1.
* 5. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumours that are refractory to standard therapy, or for which no standard therapy exists.
* 6. Has measurable disease per RECIST v1.1. that was not in a prior radiation or other locally treated area, unless imaging-based progression has been clearly documented following radiation or other local therapy

Exclusion Criteria:

* 1. Pregnant or nursing females.
* 2. Receiving concurrent anti-cancer therapy or investigational therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy).
* 3. Any remaining AEs > Grade 1 from prior anti-tumour treatment as per CTCAE v5.0, with exception of alopecia.
* 4 Subjects with primacy central nervous system (CNS) malignancy or symptomatic CNS metastases are not allowed. Subjects with asymptomatic CNS metastases are eligible if clinically controlled, which is defined as ≥4 weeks of stable neurologic function following CNS-directed therapy, and no evidence of CNS disease progression as determined by radiographic imaging ≥ 4 weeks prior to the first dose of study drug. Subjects who are receiving prednisone ≤ 10mg or equivalent steroid therapies and have a stable CNS symptom is allowed.
* 5. Subjects who have had major surgery within the 28-days from screening. If surgical procedure occurs > 28 days, they must have recovered adequately from the toxicity and/or complications from the intervention before the first dose of study drug.
* 6. Subjects with a history of tissue or organ transplantation.
* 7. Subjects who have had severe infection deemed clinically significant per Investigator within 4 weeks or signs and symptoms of any active infection within 2 weeks prior to the first dose administration.
* 8. History of human immunodeficiency virus (HIV) infection or history of autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | the first cycle of 21 days for monotherapy and the second cycle of another 21 days for combination therapy
  A DLT is defined as a toxicity occurring during the DLT observation period. Events clearly associated with the underlying disease, disease progression, a concomitant medication, or comorbidity should be excepted, and it should be considered to be at least possibly related to study drug as defined below
  Grade 5 toxicity; Grade 4 anaemia; Grade 4 thrombocytopenia lasting ≥ 7 days ; Grade 3 thrombocytopenia if associated with clinically significant bleeding (≥ Grade 2 haemorrhage) or with requirement of transfusion of platelets; Grade 4 neutropenia for ≥ 7 days ; ≥ Grade 3 neutropenia associated with infection or febrile neutropenia
Serious adverse event（SAE) | Adverse events will be collected from the time of informed consent to 90 days after the last dose or until the initiation of a new cancer treatment.
  Any SAE that is judged by the PI or designee to be related to the study medication must be reported regardless of the amount of time since the last dose received. Follow-up information collected for any initial report of an SAE must also be reported to the Sponsor within 24 hours of receipt by the PI or designee.

CONTACTS AND LOCATIONS:
Overall Officials: Prachi Bhave, M.D, Ph.D, Principal Investigator — Scientia Clinical Research Ltd
Locations (3):
- Australia (3):
  - St George Private Hospital, Kogarah
  - Blacktown Cancer and Haematology Centre, Sydney
  - Scientia Clinical Research Limited, Sydney

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD